CLINICAL TRIAL: NCT05635357
Title: Data Analysis for Drug Repurposing for Effective Alzheimer's Medicines (DREAM)- Anastrozole vs Exemestane/Letrozole
Status: Completed | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Rutgers University (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Rishi J. Desai, Assistant Professor of Medicine, Brigham and Women's Hospital
Other Study IDs: 2019P003607-11
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anastrozole: Exposure group
  Interventions: Drug: Anastrozole
- Exemestane/Letrozole: Reference group
  Interventions: Drug: Exemestane/Letrozole

INTERVENTIONS:
Drug: Anastrozole — Anastrozole claim is used as the exposure group.
  Groups: Anastrozole
Drug: Exemestane/Letrozole — Exemestane/Letrozole claim is used as the reference group.
  Groups: Exemestane/Letrozole

SUMMARY:
This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of the DREAM Study of Brigham and Women's Hospital. DREAM is led by Dr. Madhav Thambisetty, MD, PhD, Chief of the Clinical and Translational Neuroscience Section, Laboratory of Behavioral Neuroscience, National Institute on Aging (NIA) intramural research program. This study aims to evaluate the comparative risk of dementia/Alzheimer's disease onset between patients treated with medications that target specific metabolic pathways and patients treated with alternative medications for the same indication using healthcare claims data.

ELIGIBILITY:
Please see https://docs.google.com/spreadsheets/d/1GrnVsPCockqqdfxC9LWd6ndbzS2wpJVvTbCOAhn4DLM/edit?usp=sharing or Appendix A (https://drive.google.com/drive/folders/1I8FVmpPzC5wQN9DFIv1Rbwh1N0SLEv0B?usp=sharing) for full code and algorithm definitions.

Medicare timeframe: 2008 to 2018 (end of data availability)

Inclusion Criteria:

* 1. Aged >/= 65 years on the index date
* 2. Enrollment in Medicare Part A, B, and D with no HMO coverage for 365 days prior to and including cohort entry date
* 3. At least two claims with breast cancer diagnosis measured 365 days prior to drug initiation

Exclusion Criteria:

* 1. Prior history of dementia measured anytime prior to cohort entry date
* 2. Prior history of nursing home admission anytime prior to cohort entry date
* 3. Prior history of Anastrozole or Exemestane/Letrozole use anytime prior to cohort entry date

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will employ a new user, active comparator, observational cohort study design comparing Anastrozole vs Exemestane/Letrozole. The patients will be required to have continuous enrollment during the baseline period of 365 days before initiation of study drugs (cohort entry/index date). Follow-up for the outcome (dementia) differs between analyses. Follow-up begins the day after drug initiation (analysis 1, 3, 4); 180 days after drug initiation (analysis 2).
Sampling Method: Non-Probability Sample
Enrollment: 16989 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Time to dementia onset | up to 6 years
  Time to dementia onset, i.e., Alzheimer's disease, vascular dementia, senile, presenile, or unspecified dementia, or dementia in other diseases classified elsewhere. Please refer to uploaded protocol for full definition due to size limitations.

SECONDARY OUTCOMES:
Time to Alzheimer's disease onset | up to 6 years
  Time to Alzheimer's disease onset. Please refer to uploaded protocol for full definition due to size limitations.

CONTACTS AND LOCATIONS:
Overall Officials: Madhav Thambisetty, MD, PhD, Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT05635357/Prot_SAP_000.pdf